CLINICAL TRIAL: NCT02614690
Title: Is Univalving or Bivalving of Long Arm Casts for Forearm Fractures Necessary?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Mark Lee, MD, Assistant Professor of Orthopaedic Surgery, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRC118
Record Dates: First submitted 2015-05-26; First posted 2015-11-25 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Fracture of Shaft of Radius and/or Ulna; Metaphyseal Fracture of Bone of Upper Limb; Fracture of Upper Limb, Level Unspecified
Keywords: Fracture of the upper limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No split Cast of forearm fractures (Active Comparator): Patient will have a "No split cast" long arm cast applied after a closed reduction of forearm fractures. The cast will not be split. 20 patients will be randomized to this arm.
  Interventions: Procedure: No Split Cast of forearm fractures
- Univalve Split Cast of forearm fractures (Active Comparator): Patients will have a "Univalve Split Cast" long arm cast applied after undergoing closed reduction of of forearm fractures. This is a cast that is split on only one side of the cast. 20 patients will be randomized to this arm
  Interventions: Procedure: Univalve Split Cast of forearm fractures
- Bivalve Split Cast of forearm fractures (Active Comparator): Patients will have a "Bivalve Split Cast" long arm cast applied after they have undergone a closed reduction of of forearm fractures. This is a cast that will be split on both sides of the cast. 20 patients will be randomized to the bivalve split arm cast.
  Interventions: Procedure: Bivalve Split Cast of forearm fractures

INTERVENTIONS:
Procedure: No Split Cast of forearm fractures — Enroll 20 patients per arm: patients who present for long arm casts after closed reduction of forearm fractures will be randomized to one of 3 arms. Patients randomized to "No Split Cast" will have a cast that is not split, this is known as closed cast. The cast will be applied according to our Standard of Care casting. Patients will be then undergo follow-up for clinical and radiographic examinations based on the routine fracture management protocol for approximately 3 months.
  Arms: No split Cast of forearm fractures
Procedure: Univalve Split Cast of forearm fractures — Enroll 20 patients per arm: patients who present for long arm casts after closed reduction of forearm fractures will be randomized to one of 3 arms. Patients randomized to "Univalve Cast" will have a cast that is split on only one side of the cast, this is known as univalve cast. The cast will be applied according to our Standard of Care casting. Patients will be then undergo follow-up for clinical and radiographic examinations based on the routine fracture management protocol for approximately 3 months.
  Arms: Univalve Split Cast of forearm fractures
Procedure: Bivalve Split Cast of forearm fractures — Enroll 20 patients per arm: patients who present for long arm casts after closed reduction of forearm fractures will be randomized to one of 3 arms. Patients randomized to "Bivalve Cast" will have a cast that is split on both sides of the cast, this is known as bivalve cast. The cast will be applied according to our Standard of Care casting. Patients will be then undergo follow-up for clinical and radiographic examinations based on the routine fracture management protocol for approximately 3 months.
  Arms: Bivalve Split Cast of forearm fractures

SUMMARY:
This study aims to examine the need for univalve or bivalve splitting of casts in pediatric patients with forearm fractures following closed reduction and cast application in a randomized, prospective fashion.

DETAILED DESCRIPTION:
Following cast application, little is known regarding the need to split the cast, either in a univalve (a split along a single side of the cast) or bivalve (a split along both sides of the cast) fashion. Theoretically, the splitting of the cast allows for expansion and soft tissue swelling. However, review of the literature yields a paucity of evidence demonstrating the efficacy of splitting a cast. In a study by Nietosvaara et. al, a retrospective examination of 109 pediatric patients initially treated with closed cylindrical casting for closed forearm fractures were evaluated. Of these 109 patients, one-sixth required the initial cast to be split, trimmed, or removed secondary to post-traumatic swelling.

However, the splitting of a cast is not without risks in itself. Once the initial swelling dissipates, a univalved or bivalved cast can become excessively loose. This loosening has been associated with a loss of reduction. If the loss or reduction is substantial, it may require a re-reduction or operation to correct. In addition, with every use of the cast saw a patient is placed at risk for iatrogenic cast saw injury. Thermal burns and abrasions from cast saws can cause lifelong emotional and physical scars for a patient. They can also be an inciting event for litigation against the hospital and or provider, with settlements averaging greater than $12,000 per centimeter of cast saw injury.

ELIGIBILITY:
Inclusion Criteria:

* A closed isolated radial and/or ulna fracture of the forearm inclusive of metaphyseal and/or shaft level fractures.
* Forearm fractures that require closed reduction (with or without conscious sedation)
* Patients between the ages of 3 and 12 years old

Exclusion Criteria:

1. Specific exclusions

   * Age less than 3 or greater than 12
   * Patients presenting with an associated neurological or vascular injury caused by the fracture
   * Patients presenting with an open fracture
   * Patients requiring operative treatment following the initial fracture evaluation
   * Ipsilateral upper extremity fracture
   * Patients intubated or with a pre-existing condition that prevents them from verbalizing symptoms of discomfort
2. Generic exclusion: "Subjects not meeting all inclusion criteria."

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lee, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing individual data. Plan is to publish the data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients between ages 3 to 13 with closed shaft or distal third radius and ulna fracture requiring reduction were enrolled at Connecticut Children's Medical Center Emergency room between 2013 and 2015.
Pre-assignment Details: There were no pre-assignment details.
Period: Overall Study
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.6 (3.818376618) | 8.1 (5.515432893) | 9.0 (4.737615434) | 8.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 4 | 6 | 8 | 18
  Sex: Male | 16 | 14 | 12 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Complication Rate of the Cast Type
Description: This data will be able to help physicians and ER personnel help this patient population with the least number of cast complications and therefore allow for a more efficient use of resources since cast modifications could be minimized. Metrics used to characterize complications are the radiographic union used to determine speed of healing and the number of unplanned ER or clinic visits for cast modifications.
Time Frame: <60 days corresponding to total study time and consistent with outcome 6
Measure: Number; unit: participants
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
participants | 9 | 12 | 8

2. Other Pre Specified Outcome: Cast Index
Description: The cast index is a measure of potential for cast failure described by Chess et al. in 1994. The cast index is calculated as the sagittal width measure divided by the coronal cast width measure at the fracture site. A ratio between these measures of 0.7 or greater for pediatric forearms is considered acceptable. For each patient in this study the cast index was calculated as described above. The average cast index for each of the 3 groups was then presented as the final result.
Time Frame: Immediately after cast application (<1 day)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
ratio | .88 (0.11) | .90 (0.09) | .83 (0.05)

3. Other Pre Specified Outcome: Number of Participants With Different Fracture Characteristics
Time Frame: Less than 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
Participants
  Distal Radius/Ulna | 10 | 8 | 13
  Distal Third Radius/Ulna | 5 | 4 | 5
  Midshaft Radius/Ulna | 3 | 6 | 2
  Proximal Third Radius/Ulna | 2 | 2 | 0

4. Other Pre Specified Outcome: Pain Levels
Description: Pain levels were assessed using the validated Wong-Baker FACES visual pain rating scale. This scale presents a total of 6 options for pain- none, 1, 2, 3, 4, and 5- with 5 corresponding to the greatest amount of pain. During the analysis it was decided to group these into 5 categories: No pain which was equal to those selecting none, Mild corresponding to those selecting 1, Moderate pain corresponding to those that selected either 2 or 3, and Severe pain corresponding to those that selected either 4 or 5. Patients with no response were placed into the group "no response".
Time Frame: one week
Measure: Count of Participants; unit: Participants
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
Participants
  No pain | 12 | 9 | 12
  Mild Pain | 2 | 0 | 3
  Moderate pain | 2 | 5 | 1
  Severe pain | 1 | 3 | 3
  No response | 3 | 3 | 1

5. Other Pre Specified Outcome: Number of Patients With Different Fracture Treatments
Time Frame: 4 weeks
Measure: Number; unit: participants
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
participants
  Wedge for loss of reduction | 4 | 10 | 6
  Surgical stabilization | 0 | 1 | 0

6. Other Pre Specified Outcome: Number of Participants With Different Cast Complications
Time Frame: Day 1 to day 56
Measure: Number; unit: participants
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
participants
  Compartment syndrome | 0 | 0 | 0
  Cast saw abrasions | 0 | 0 | 0
  Unplanned Office Visits | 2 | 1 | 1
  Unplanned Cast Modifications Visits | 3 | 0 | 1
  Surgical Stablization | 0 | 1 | 0
  Cast Wedged | 4 | 10 | 6

7. Other Pre Specified Outcome: Average Time for First Follow-up Appointment
Description: Average time from reduction and casting to the first follow-up visit.
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
Number analyzed (Participants) | 20 | 20 | 20
days | 5.9 (2.1) | 6.4 (1.7) | 5.8 (2.3)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected 5 to 10 days, and 6 weeks after the initial cast application. Also captured at visit that occurred at the discretion of the provider.
Arm/Group | No Split Cast of Forearm Fractures | Univalve Split Cast of Forearm Fractures | Bivalve Split Cast of Forearm Fractures
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The study was powered to detect a two patient difference in the incidence of cast related compartment syndrome and neurologic injuries between the three casting groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No